CLINICAL TRIAL: NCT04748705
Title: A Double-Blinded, Randomized, Placebo-Controlled, Phase 2B Trial of IMC-1 for the Treatment of Fibromyalgia
Brief Title: Fibromyalgia Outcome Research Trial Evaluating Synergistic Suppression of HSV-1
Acronym: FORTRESS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Virios Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PRID-202
Record Dates: First submitted 2021-02-05; First posted 2021-02-10 (Actual); Last update posted 2022-09-27 (Actual); Status verified 2022-09

CONDITIONS: Fibromyalgia
Keywords: Pain
MeSH Terms: conditions — Fibromyalgia; Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- IMC-1 Oral Tablet (Experimental): 2X IMC-1 Tablet taken orally, each morning and evening.
  Interventions: Drug: IMC-1
- Placebo (Placebo Comparator): 2X Placebo Tablet taken orally, each morning and evening.
  Interventions: Drug: Placebo BID Tablet

INTERVENTIONS:
Drug: IMC-1 — Patients will take 1 tablet twice daily, each morning and evening, of randomly assigned study drug orally starting on Day 1 through study duration.
  Arms: IMC-1 Oral Tablet
Drug: Placebo BID Tablet — Patients will take 1 tablet twice daily, each morning and evening, of randomly assigned study drug orally starting on Day 1 through study duration.
  Arms: Placebo

SUMMARY:
Randomized, double-blind, placebo-controlled, 16-week study designed to explore the safety and efficacy of IMC-1 for the treatment of patients with fibromyalgia.

ELIGIBILITY:
Inclusion Criteria:

* The patient is female, 18 to 65 years of age, inclusive.
* The patient has a diagnosis of primary FM as defined by the 2016 Revisions to the 2010/2011 fibromyalgia diagnostic criteria (American College of Rheumatology Preliminary Diagnostic Criteria)
* The in clinic 7-day recall VAS scale average daily pain intensity score at Screening visit within protocol defined range.

Exclusion Criteria:

* Any underlying medical or psychiatric condition that could impact their safe participation per protocol.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 422 (Actual)
Dates: Start 2021-06-03 (Actual); Primary Completion 2022-08-05 (Actual); Study Completion 2022-08-05 (Actual)

PRIMARY OUTCOMES:
Mean Pain Score | 16 Week
  Change from Baseline to Week 16 endpoint in the diary Numerical Rating Scale (NRS) weekly average of daily self-reported average pain severity scores. Scores range from 0 to 10 where a higher score means worse outcome.

CONTACTS AND LOCATIONS:
Locations (42):
- United States (42):
  - IMC Study Site, Birmingham, Alabama
  - IMC Study Site, Rogers, Arkansas
  - IMC Study Site, Oceanside, California
  - IMC Study Site, Riverside, California
  - IMC Study Site, Sacramento, California
  - IMC Study Site, San Diego, California
  - IMC Study Site, Santa Ana, California
  - IMC Study Site, Temecula, California
  - IMC Study Site, Jacksonville, Florida
  - IMC Study Site, Ocala, Florida
  - IMC Study Site, Oldsmar, Florida
  - IMC Study Site, Orlando, Florida
  - IMC Study Site, Tampa, Florida
  - IMC Study Site, Alpharetta, Georgia
  - IMC Study Site, Gurnee, Illinois
  - IMC Study Site, Evansville, Indiana
  - IMC Study Site, Des Moines, Iowa
  - IMC Study SIte, Prairie Village, Kansas
  - IMC Study Site, Covington, Louisiana
  - IMC Study Site, New Orleans, Louisiana
  - IMC Study Site, Prairieville, Louisiana
  - IMC Study Site, Boston, Massachusetts
  - IMC Study Site, North Dartmouth, Massachusetts
  - IMC Study Site, Jackson, Mississippi
  - IMC Study Site, Las Vegas, Nevada
  - IMC Study Site, Albuquerque, New Mexico
  - IMC Study Site, Cedarhurst, New York
  - IMC Study Site, Williamsville, New York
  - IMC Study Site, Cincinnati, Ohio
  - IMC Study Site, North Canton, Ohio
  - IMC Study Site, Oklahoma City, Oklahoma
  - IMC Study Site, Tulsa, Oklahoma
  - IMC Study Site, Portland, Oregon
  - IMC Study Site, Allentown, Pennsylvania
  - IMC Study Site, Warwick, Rhode Island
  - IMC Study Site, Chattanooga, Tennessee
  - IMC Study Site, Knoxville, Tennessee
  - IMC Study Site, Austin, Texas
  - IMC Study Site, Dallas, Texas
  - IMC Study Site, Salt Lake City, Utah
  - IMC Study Site, Charlottesville, Virginia
  - IMC Study Site, Everett, Washington

IPD SHARING:
Plan to Share IPD: No
No: There is not a plan to make IPD available.

REFERENCES:
- [Background] Pridgen WL, Duffy C, Gendreau JF, Gendreau RM. A famciclovir + celecoxib combination treatment is safe and efficacious in the treatment of fibromyalgia. J Pain Res. 2017 Feb 22;10:451-460. doi: 10.2147/JPR.S127288. eCollection 2017. PMID 28260944